CLINICAL TRIAL: NCT01595971
Title: Distance Education Versus Usual Care in the Qualification of Asthma Care: A Cluster Randomized Clinical Trial - RESPIRANET
Brief Title: Distance Education Versus Usual Care Qualification in Asthma Care
Acronym: RESPIRANET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MED/FNS 774/08
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Continuing education; Primary health care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuing education (Experimental): RESPIRANET is a multifaceted intervention directed at professionals of the Family Health Teams in the inner cities.Includes telemedicine, reminders, video conferences, educational materials for patients and consultants.
  Interventions: Behavioral: Continuing education
- Usual Care (Placebo Comparator): usual care
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: Continuing education — Includes telemedicine, reminders, video conferences, educational materials for patients and consultants.
  Other Names: RESPIRANET
  Arms: continuing education
Other: usual care — Received the usual care provided
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of multifaceted educational interventions in the care of asthma, conducted remotely over the platform TelessaúdeRS in teams of the Family Health Strategy and the consequent clinical improvement patients.

DETAILED DESCRIPTION:
Cluster-randomized trial with follow-up of 6 months. The aim of this study is to determine whether multifaceted interventions performed at a distance for the care of asthma symptoms reduce overhead, improve asthma control and qualify the care provided to patients.

ELIGIBILITY:
Inclusion Criteria:

* Practice:Participate in the Telessaúde/RS. Minimal staff consisting of a general practitioner, nurse, nurse and community health agents (CHA), ability to give at least ten patients diagnosed with asthma, located in a municipality to make available for free inhaled medication (short-acting bronchodilators and corticosteroids ) for the treatment of asthma and willingness to participate in the study.
* Patients: 5 to 45 years with a diagnosis of asthma made by a physician and register at least one consultation for asthma or an asthma-related hospitalization during the year preceding the beginning of the study.

Exclusion Criteria:

* Patients with other chronic diseases with pulmonary complications such as tuberculosis, cancer and cystic fibrosis or those with severe mental illness

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 467 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2011-12-16 (Actual); Study Completion 2011-12-16 (Actual)

PRIMARY OUTCOMES:
Symptom burden, measured as the number of self-reported asthma symptom days (ASD). ASD is based on 2 week recall. | six months
  The definition of a symptom day includes presence of any of the four types of asthma symptoms: wheeze, cough, night time awakening ou shortness of breath. The results will be collected through the application of standardized questionnaires.

SECONDARY OUTCOMES:
Asthma control | 6 months
  Control of asthma will be evaluated by the excessive use of relief medication in the last month.
Health care utilization | 6 meses
  Proportion of unscheduled medical visits during the follow-up
Proportion of patients in use inhaled corticosteroids | 6 meses
  Use of inhaled corticosteroids assessed by the proportion of patients who require medication to prevent asthma symptoms that are in use of inhaled corticosteroids.

CONTACTS AND LOCATIONS:
Overall Officials: Erno Harzheim, PHD, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Collaborator website — http://www.ufrgs.br/telessauders